CLINICAL TRIAL: NCT01169077
Title: A Phase I, Randomized, Controlled Dosage-Escalation Study of the Safety and Reactogenicity of the EP1300 Polyepitope DNA Vaccine Against Plasmodium Falciparum Malaria Administered Via Electroporation to Healthy Adults
Brief Title: EP1300 Polyepitope DNA Vaccine Against Plasmodium Falciparum Malaria
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 08-0008; N01AI80005C
Record Dates: First submitted 2010-07-22; First posted 2010-07-23 (Estimated); Last update posted 2012-11-16 (Estimated); Status verified 2012-11

CONDITIONS: Plasmodium Falciparum Malaria
Keywords: malaria, plasmodium falciparum, electroporation
MeSH Terms: conditions — Malaria, Falciparum; Malaria

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- Group I: 0.25 mg EP-1300 (Experimental): Ten subjects will receive 3 immunizations of EP1300, 0.25 mg, on Day 0, Day 28 and Day 56. Three control subjects in this group will receive placebo injections at the same timepoints.
  Interventions: Drug: Placebo; Biological: EP-1300
- Group II: 1.0 mg EP-1300 (Experimental): Ten subjects will receive 3 immunizations of EP1300, 1.0 mg, on Day 0, Day 28 and Day 56. Three control subjects in this group will receive placebo injections at the same timepoints.
  Interventions: Drug: Placebo; Biological: EP-1300
- Group III: 4.0 mg EP-1300 (Experimental): Ten subjects will receive 3 immunizations of EP1300, 4.0 mg, Day 0, Day 28 and Day 56. Three control subjects in this group will receive placebo injections at the same timepoints.
  Interventions: Drug: Placebo; Biological: EP-1300

INTERVENTIONS:
Drug: Placebo — Injections of normal saline to be used as control; given at Days 0, 28, and 56. Administered via electroporation, using a DNA vaccine delivery device, in the deltoid.
Biological: EP-1300 — Single DNA plasmid dissolved in phosphate-buffered saline (PBS). Dose levels: 0.25, 1 and 4 mg based on DNA content, administered on Days 0, 28 and 56 via electroporation using a DNA vaccine delivery device, in the deltoid.

SUMMARY:
Malaria, a disease responsible for over one million deaths per year, is caused by a germ spread by mosquito bites. The purpose of this study is to evaluate a vaccine designed for the prevention of malaria caused by the parasite, Plasmodium falciparum, and to evaluate the device used to give the vaccine. This study will provide information on how safe, effective, and tolerable the vaccine is in healthy adults. The participants will be assigned, by chance, to receive 3 doses/shots of the vaccine or a placebo (substance that contains no medication) by injection in the upper arm. Study participants will include 39 healthy adults aged 18-40 years who have not been exposed to malaria and who will enroll at the Emory Vaccine and Treatment Evaluation Unit in Atlanta, Georgia. Study procedures include physical exams and several blood samples. Participants will be involved in the study for approximately seven and one half months.

DETAILED DESCRIPTION:
Malaria is a mosquito-borne disease caused by protozoan parasites of the genus Plasmodium (P.). It is estimated that there are 350-500 million clinical cases of malaria per year, accounting for over one million deaths. The majority of deaths occur among children under five years of age in Africa, especially in those areas with poor access to healthcare services. Severe disease occurs most frequently with P. falciparum, at least partially due to its ability to infect a higher percentage of erythrocytes and to adhere to capillary walls. Development of a safe and effective vaccine targeting P. falciparum is a major public health goal. To be truly effective in the general population, a vaccine should induce responses targeting "immunologically" conserved regions. Epitope-based vaccines represent a very logical approach to this problem because they can be designed to focus immune responses only on conserved epitopes. The proposed clinical trial will be the first to evaluate a novel deoxyribonucleic acid (DNA)-based, polyepitope vaccine against P. falciparum malaria. The study will be conducted as a phase I, randomized, prospective, controlled, single-center, dose-escalating trial. This study is designed to provide information regarding the safety and tolerability of the EP (Electroporation) 1300 vaccine that will allow further development of the vaccine in future studies. Immunogenicity will be assessed in a preliminary fashion as a secondary endpoint. The primary objective of this study is to evaluate the safety, reactogenicity and tolerability of the EP1300 (DNA) vaccine administered via electroporation in healthy adult volunteers. The secondary objectives are to obtain preliminary immunogenicity data for the EP1300 polyepitope DNA vaccine as assessed by interferon-gamma enzyme-linked immunospot assay and to assess the tolerability of the administration procedure in healthy volunteers. Thirty-nine healthy adults aged 18 through 40 who have no previous history of malaria exposure or infection, no history of travel to malaria-endemic areas, and who have not received vaccines for malaria infection will be enrolled in this study. Subjects will be randomized to receive 3 doses of either the DNA vaccine or normal saline placebo at day 0, 28, and 56. DNA doses will be administered in dose-escalating fashion from 0.25 mg to 4 mg. Dose escalation will proceed following a review of all safety data up to and including the 2-week safety data time point following the second immunization in the prior dosage group; review includes participation by Division of Microbiology and Infectious Diseases and the Safety Monitoring Committee.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, 18 through 40 years old, who deny exposure to or infection with malaria or prior participation in a malaria vaccine study.
* In good health, defined as a person who consents to participate in the trial, agrees to not donate blood until 6 months following the last blood draw in the protocol, and whose clinical laboratory assessments are within parameters as specified in this protocol in Appendix C, (Acceptable Screening Laboratory Ranges). (Women of childbearing potential (not surgically sterile or postmenopausal for >/= 1 year) must not be pregnant as indicated by a negative pregnancy test (urine or serum) within 24 hours prior to vaccine administration.
* Women of childbearing potential who are at risk of becoming pregnant must agree to practice adequate contraception (i.e., barrier methods in conjunction with spermicidal gel, abstinence, monogamous relationship with vasectomized partner, intrauterine devices, Depo-Provera, Norplant, oral contraceptives, contraceptive patches or other licensed, effective methods) until 30 days following receipt of the last dose of vaccine.
* Able to understand and comply with planned study procedures.
* Able to provide informed consent prior to initiation of any study procedures and be available for all study visits.
* Have access to a telephone.

Exclusion Criteria:

* Prior history of travel to a malaria-endemic area.
* History of previous malaria infection.
* Planned travel to a malaria-endemic area during the course of the study.
* History of splenectomy.
* Known hypersensitivity to components of the vaccine (deoxyribonucleic acid, phosphate-buffered saline, potassium dihydrogen phosphate, sodium hydrogen phosphate) or to kanamycin or other aminoglycoside antibiotics.
* Is female of child-bearing potential who is breastfeeding or intends to become pregnant during the study period up to 30 days following receipt of the last dose of vaccine.
* Has immunosuppression as a result of an underlying illness or treatment with immunosuppressive or cytotoxic drugs, or use of anticancer radiation therapy within the preceding 60 months.
* History of significant cardiac abnormality and/or abnormal baseline electrocardiogram (ECG) readout, and/or history of arrhythmia, including any cardiac pre-excitation syndromes (such as Wolff Parkinson White) or other cardiac syndromes or diseases (such as congestive heart failure) associated with arrhythmias, a history of syncopal episodes, and/or family history of prolonged QTc syndrome.
* Subjects with a seizure disorder, except for those who have been seizure free for 5 years or are felt to be at low risk for seizure as determined by their neurologist (the effects of electric field generation near sites where the threshold of field sensitivity is low is unknown).
* Subjects with hemophilia, thrombocytopenia, bleeding or clotting disorders, muscular atrophy or muscular/neuromuscular degenerative disorders.
* Presence of any implanted any electronic stimulation device, such as cardiac demand pacemakers, automatic implantable cardiac defibrillator, nerve stimulators, or deep brain stimulators.
* Individuals in which a skin-fold measurement of the cutaneous and subcutaneous tissue for all eligible injection sites (deltoid muscles with intact lymph drainage) exceeds 40 millimeters.
* Presence of surgical or traumatic metal implant in the upper limb and/or upper torso.
* Subjects with tattoos, lesions, rashes, scars or tumors at the proposed sites of administration.
* Has an active neoplastic disease (excluding non-melanoma skin cancer or prostate cancer that is stable in the absence of therapy) or a history of any hematologic malignancy. Active is defined as: no neoplastic disease or treatment for neoplastic disease within the past 5 years.
* Has long-term use (greater than 2 weeks) of oral or parenteral steroids, or high-dose inhaled steroids (greater than 800 micrograms per day of beclomethasone dipropionate or equivalent) within the preceding 6 months (nasal and topical steroids are allowed).
* Has a history of receiving immunoglobulin or other blood products within the 3 months prior to enrollment in this study.
* Has received any other licensed vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to enrollment in this study, or plans to receive any other licensed vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) following each study vaccination.
* Has an acute or chronic medical condition that, in the opinion of the investigator, would render vaccination unsafe or would interfere with the evaluation of responses (this includes, but is not limited to: known cardiac arrhythmia or coronary artery disease, known chronic liver disease, significant renal disease, unstable or progressive neurological disorders, diabetes mellitus, and transplant recipients, bleeding disorders, or skin conditions, e.g. psoriasis).
* Has a history of severe reactions suggesting anaphylaxis following any previous vaccination.
* Has an acute illness or has an oral temperature greater than 99.9 degrees Fahrenheit (37.7 degrees Celsius) within 3 days prior to enrollment.
* Has received an experimental agent (vaccine, drug, biologic, device, blood product, or medication) within 1 month prior to enrollment in this study, or expect to receive an experimental agent during the study period.
* Has any condition that would, in the opinion of the site principal investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.
* Has a diagnosis of schizophrenia, bipolar disease or other severe (disabling) chronic psychiatric diagnosis.
* Has been hospitalized for psychiatric illness, history of suicide attempt or confinement for danger to self or others.
* Is receiving psychiatric drugs (aripiprazole, clozapine, ziprasidone, haloperidol, molindone, loxapine, thioridazine, thiothixene, pimozide, fluphenazine, risperidone, mesoridazine, quetiapine, trifluoperazine, trifluopromazine, chlorprothixene, chlorpromazine, perphenazine, olanzapine, carbamazepine, divalproex sodium, lithium carbonate or lithium citrate). Subjects who are receiving a single antidepressant drug and are stable for at least 3 months prior to enrollment without decompensating are allowed enrollment into the study.
* Positive serology for human immunodeficiency virus, hepatitis B, or hepatitis C infection.
* Abnormal values on clinical safety laboratory tests obtained during screening.
* Has a history of alcohol or drug abuse in the 5 years prior to enrollment.
* Has a history of Guillain-Barré syndrome.
* Has any condition that the investigator believes may interfere with successful completion of the study.
* Plans to enroll in another clinical trial at any time during the study period.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2010-08; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
The number of serious adverse events considered associated with the vaccine. | Reported at any point during follow-up.
The number of subjects reporting solicited systemic adverse events of severity (grade 3) or higher. | Within 14 days after receiving any dose of vaccine.
The number of subjects experiencing spontaneous adverse events of severity (grade 3) or higher and considered associated with the vaccine. | Reported at any point during follow-up.
The number of subjects reporting local reactogenicity of severity (grade 3) or higher. | Within 14 days after receiving any dose of vaccine.

SECONDARY OUTCOMES:
Responses to tolerability questionnaire used to document subject feedback of electroporation mediated DNA vaccine delivery; proportion of subjects judging the procedure to be suitable for use in context of a prophylactic malaria vaccine. | Day 0, 28 and 56.
Antibody titers in serum measured against malaria circumsporozoite protein [Geometric Mean Titer and individual log Enzyme-Linked Immunosorbent Assay (ELISA) units] for subjects in groups II and III. | Day 0, 42, and 70.
Sample number showing positive falciparum-specific responses, Geometric Mean Titer spot-forming cells/million peripheral blood mononuclear cell per cohort, subject frequency per cohort with at least 1 positive response. | Days 0, 42 and 70.
Interferon-gamma Enzyme-Linked Immunospot Assay (ELISPOT) assay. | Days 0, 42 and 70.

CONTACTS AND LOCATIONS:
Locations (1):
- Emory Children's Center - Pediatric Infectious Diseases, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Spearman P, Mulligan M, Anderson EJ, Shane AL, Stephens K, Gibson T, Hartwell B, Hannaman D, Watson NL, Singh K. A phase 1, randomized, controlled dose-escalation study of EP-1300 polyepitope DNA vaccine against Plasmodium falciparum malaria administered via electroporation. Vaccine. 2016 Nov 4;34(46):5571-5578. doi: 10.1016/j.vaccine.2016.09.041. Epub 2016 Sep 30. PMID 27697302